CLINICAL TRIAL: NCT02517021
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Control Study to Evaluate the Safety and Efficacy of IV Pro-netupitant/Palonosetron (260 mg/0.25 mg) Combination for the Prevention of Chemotherapy-induced Nausea and Vomiting in Repeated Chemotherapy Cycles in Patients Receiving Highly Emetogenic Chemotherapy
Brief Title: A Safety Study of Intravenous Pro-Netupitant and Palonosetron Combination for the Prevention of Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: PSI CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NEPA-15-18
Record Dates: First submitted 2015-08-03; First posted 2015-08-06 (Estimated); Results first posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Palonosetron; netupitant, palosentron drug combination; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pro-netupitant/Palonosetron plus Dexamethasone (Experimental): Intravenous Pro-netupitant/Palonosetron (260 mg/0.25 mg) powder for solution for infusion (on Day 1) with oral dexamethasone prior to each scheduled chemotherapy cycle
  Interventions: Drug: Pro-netupitant/Palonosetron; Drug: Dexamethasone
- Netupitant/Palonosetron plus Dexamethasone (Active Comparator): Oral netupitant/palonosetron (300 mg/0.50 mg) hard capsule (on Day 1) with oral dexamethasone prior to each scheduled chemotherapy cycle
  Interventions: Drug: Netupitant/Palonosetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pro-netupitant/Palonosetron
  Other Names: IV NEPA FDC
  Arms: Pro-netupitant/Palonosetron plus Dexamethasone
Drug: Netupitant/Palonosetron
  Other Names: Oral NEPA FDC
  Arms: Netupitant/Palonosetron plus Dexamethasone
Drug: Dexamethasone

SUMMARY:
NEPA-15-18 is a clinical study assessing safety of pro-netupitant and palonosetron, two antiemetic drugs, given with oral dexamethasone. The objective of the study is to evaluate if pro-netupitant and palonosetron are safe when administered to prevent nausea and vomiting after administration of repeated cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Cycle 1

* Signed written informed consent
* Histologically or cytologically confirmed solid tumor malignancy.
* Naïve to cytotoxic chemotherapy. Previous biological or hormonal therapy will be permitted.
* Scheduled to receive at least 4 repeated consecutive cycles of the following highly emetogenic reference chemotherapies (HEC), alone or in combination with other chemotherapeutic agents on Day 1: cisplatin administered as a single IV dose of ≥ 70 mg/m2; cyclophosphamide ≥1500 mg/m2; carmustine (BCNU) >250mg/m2; dacarbazine (DTIC); mechloretamine (nitrogen mustard)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2 .
* If a patient is female, she shall be of non-childbearing potential or of childbearing potential using reliable contraceptive measures and having a negative urine pregnancy test.
* Hematologic and metabolic status adequate for receiving an highly emetogenic regimen based on laboratory criteria (Total Neutrophils,Platelets, Bilirubin, Liver enzymes, Serum Creatinine or Creatinine Clearance)
* Able to read, understand, follow the study procedure and complete patient diary.

Cycles 2 to 4:

The following inclusion criteria must be checked prior to inclusion at each repeated cycle:

* Participation in the study during the next cycle of chemotherapy is considered appropriate by the Investigator and does not pose unwarranted risk to the patient.
* Scheduled to receive the same chemotherapy regimen as Cycle 1 or one of the reference chemotherapies as defined in Inclusion criterion 5 for Cycle 1.
* If a patient is female, she shall be of non--childbearing potential or of childbearing potential using reliable contraceptive measures and having a negative urine pregnancy test.
* Adequate hematologic and metabolic status according to the Investigator's opinion.

Exclusion Criteria:

Cycle 1

* Lactating woman.
* Active infection or uncontrolled disease except for malignancy that may pose unwarranted risks in administering the study drugs to the patient.
* Current use of illicit drugs or current evidence of alcohol abuse.
* Scheduled to receive moderately or highly emetogenic chemotherapies from Day 2 to Day 5.
* Received or is scheduled to receive radiation therapy to the abdomen or the pelvis within 1 week prior to the start of the reference chemotherapy administration on Day 1 or between Days 1 to 5.
* Any vomiting, retching, or nausea (grade ≥ 1 as defined by National Cancer Institute) within 24 hours prior to the start of the reference chemotherapy administration on Day 1.
* Symptomatic primary or metastatic CNS malignancy.
* Known hypersensitivity or contraindication to 5-HT3 receptor antagonists, to dexamethasone or to NK-1 receptor antagonists.
* Known contraindication to the IV administration of 50 mL 5% glucose solution.
* Previously received an NK-1 receptor antagonist.
* Participation in a previous clinical trial involving IV pro-netupitant or oral netupitant administered alone or in combination with palonosetron.
* Any investigational drugs (other than those given in this study) taken within 4 weeks prior to Day 1, and/or is scheduled to receive any investigational drug during the present study.
* Systemic corticosteroid therapy at any dose within 72 hours prior to the start of reference chemotherapy administration on Day 1. Topical and inhaled corticosteroids are permitted.
* Scheduled to receive bone marrow transplantation and/or stem cell rescue therapy.
* Scheduled to receive any strong or moderate inhibitor of CYP3A4 or its intake within 1 week prior to Day 1.
* Scheduled to receive any of the following CYP3A4 substrates within 1 week prior to Day 1: terfenadine, cisapride, astemizole, pimozide.
* Received within 4 weeks prior to Day 1 or scheduled to receive any CYP3A4 inducer.
* Any medication with known or potential antiemetic activity within 24 hours prior to the start of reference chemotherapy administration on Day 1 of Cycle 1, including but not limited to 5-HT3 receptor antagonists and NK-1 receptor antagonists
* History or predisposition to cardiac conduction abnormalities, except for incomplete right bundle branch block
* History of Torsade de Point or known history of risk factors for Torsade de Point (heart failure, hypokalemia, family history of Long QT Syndrome).
* Severe cardiovascular diseases diagnosed within 3 months prior to Day 1 of first cycle, including myocardial infarction, unstable angina pectoris, significant valvular or pericardial disease, history of ventricular tachycardia, symptomatic Congestive Heart Failure (CHF) New York Heart Association (NYHA) class III-IV, and severe uncontrolled arterial hypertension.
* Any illness or condition that, in the opinion of the Investigator, may confound the results of the study or pose unwarranted risks in administering the investigational product to the patient.
* Concurrent medical condition that would preclude administration of dexamethasone such as systemic fungal infection or uncontrolled diabetes.

Cycles 2 to 4:

The following exclusion criteria must be checked prior to inclusion in each repeated cycle:

* Lactating woman.
* Active infection or uncontrolled disease except for malignancy that may pose unwarranted risks in administering the study drugs to the patient.
* Started any of the restricted medications.
* Any vomiting, retching, or nausea (grade ≥ 1 as defined by National Cancer Institute) within 24 hours prior to the start of reference chemotherapy administration on Day 1.
* Received or is scheduled to receive radiation therapy to the abdomen or the pelvis within 1 week prior to the start of the reference chemotherapy administration on Day 1 or between Days 1 to 5.
* Symptomatic primary or metastatic CNS malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (11):
  - Sarcoma Oncology Center, Santa Monica, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - St. Mary's Medical Center, Grand Junction, Colorado
  - Well Pharma Medical Research Corporation, Miami, Florida
  - Illinois CancerCare, Peoria, Illinois
  - Indiana University Health Bloomington, Bloomington, Indiana
  - Christus St. Frances Cabrini Hospital, Alexandria, Louisiana
  - North Shore Hematology Oncology Associates PC, East Setauket, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - West Cancer Center, Germantown, Tennessee
  - Provision Center for Biomedical Research, Knoxville, Tennessee
- Austria (5):
  - University Hospital Graz, Department of Internal Medicine, Graz
  - Krems Country Hospital, Krems
  - Hospital Elisabethinen Linz GmbH, Internal Department #1 - Hemato-Oncology, Linz
  - General Hospital Linz GmbH, Internal Medicine Department #3 - Center for Hematology and Medical Oncology, Linz
  - University Hospital St. Poelten,1st Medical Department, Sankt Pölten
- Croatia (4):
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Center "Sestre milosrdnice", Zagreb
  - University Hospital Centre Zagreb "Jordanovac", Zagreb
- Czechia (6):
  - University Hospital Brno. Clinic of Pulmonary Diseases and Tuberculosis, Brno
  - University Hospital, Brno
  - Hospital Novy Jicin, Department of Oncology, Nový Jičín
  - Thomayer's Hospital, Clinic of Pneumology, Prague
  - Hospital Na Bulovce, Prague
  - Masaryk's Hospital Usti nad Labem, Oncology Dept, Ústí nad Labem
- Germany (5):
  - Onkoligische Schwerpunktpraxis Bielefeld, Bielefeld
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - Hannover Medical School, Hanover
  - Universitaetsklinikum Leipzig; Universitaeres Krebszentrum (UCCL), Leipzig
  - Staedtisches Klinikum Muenchen GmbH; Klinikum N euperlach, München
- Israel (3):
  - Barziali Medical Center, Oncology Unit, Ashkelon
  - Soroka University Medical Center,Oncology division, Beersheba
  - Rambam Health Care Campus, Haifa
- Italy (6):
  - S. G. Moscati Hospital, Medical Oncology Division, Avellino
  - cientific Institute of Romagna for the Study and Treatment of Cancer (IRST), IRCCS, Meldola
  - National Cancer Institute, IRCCS, Medical Oncology Department, Milan
  - Azienda Socio Sanitaria Territoriale-Monza (ASST-Monza) - Oncology Department, Monza
  - Regional Hospital "San Carlo", Potenza
  - Local Healthcare Company of Vimercate (ASST Vimercate), Vimercate
- Poland (7):
  - Provincial Hospitals in Gdynia Sp. z o.o. (LLC), Gdynia
  - Lord's Transfiguration Teaching Hospital, Department of Chemotherapy, Poznan
  - Specialist Hospital in Prabuty Sp. z o .o. (LLC), Department of Pulmonology, Prabuty
  - Zofia Zamoyska nee Tarnowska Provincial Hospital in Tarnobrzeg, Tarnobrzeg
  - Ludwik Rydygier Provincial Hospital, Torun
  - Maria Sklodowska-Curie Institute of Oncology, Department of Lung and Thoracic Cancers, Warsaw
  - MAGODENT Sp. z o .o. (LLC), Branch No. 4, Department of Clinical Oncology/Chemotherapy, Warsaw
- Serbia (6):
  - Clinical Center of Serbia, Clinic of Pulmonology, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Clinic of Oncology, Belgrade
  - Institute of Oncology and Radiology of Serbia, Clinic of Medical Oncology, Belgrade
  - Military Medical Academy, Belgrade
  - Institute of Pulmonary Diseases of Vojvodina, Pulmonary Oncology Clinic, Kamenitz
  - Oncology Institute of Vojvodina, Kamenitz
- South Africa (2):
  - GVI Outeniqua Oncology Unit, George
  - Medical Oncology Centre of Rosebank, Johannesburg
- Spain (5):
  - Hospital Nuestra Senora de Valme, Seville, Andalusia
  - Our Lady of Sonsoles Hospital, Ávila
  - Hospital Puerta de Hierro, Madrid
  - Hospital La Paz, Oncology Department, Madrid
  - University Hospital Quiron Madrid, Department of Oncology, Madrid
- Ukraine (14):
  - Chernivtsi Regional Clinical Oncology Center, Day Care Unit, Chernivtsi
  - Clinical Oncology Center, Department of Chemotherapy, Dnipropetrovsk
  - Dnipropetrovsk City Multispecialty Clinical Hospital #4, Department of Chemotherapy, Dnipropetrovsk
  - Regional Clinical Oncology Center, Chemotherapy Department, Ivano-Frankivsk
  - S.P. Hryhoriev Institute of Medical Radiology, Department of Chemotherapy, Kharkiv
  - Kharkiv Regional Clinical Oncology Center, Chemotherapy Department #1, Kharkiv
  - Khmelnytskyi Regional Oncology Center, Surgery Department #1, Khmelnytskyi
  - Kryvyi Rih Oncology Center, Department of Chemotherapy, Kryvyi Rih
  - Lviv State Regional Treatment and Diagnostics Oncology Center, Department of Chemotherapy, Lviv
  - Ternopil Regional Public Clinical Oncology Center, Ternopil
  - LTD UNIMED Adjara, Uzhhorod
  - Zakarpattia Regional Clinical Oncology Center, Department of Chemotherapy, Uzhhorod
  - Vinnytsia Regional Clinical Oncology Center, Department of Chemotherapy, Vinnytsia
  - Zaporizhia Regional Clinical Oncology Center, Thoracic Department, Zaporizhia

REFERENCES:
- [Derived] Schwartzberg L, Roeland E, Andric Z, Kowalski D, Radic J, Voisin D, Rizzi G, Navari R, Gralla RJ, Karthaus M. Phase III safety study of intravenous NEPA: a novel fixed antiemetic combination of fosnetupitant and palonosetron in patients receiving highly emetogenic chemotherapy. Ann Oncol. 2018 Jul 1;29(7):1535-1540. doi: 10.1093/annonc/mdy169. PMID 29722791

RESULTS

PARTICIPANT FLOW:
Groups:
- Pro-netupitant/Palonosetron Plus Dexamethasone: Intravenous Pro-netupitant/Palonosetron (260 mg/0.25 mg) powder for solution for infusion (on Day 1) with oral dexamethasone prior to each scheduled chemotherapy cycle
  Pro-netupitant/Palonosetron
  Dexamethasone
- Netupitant/Palonosetron Plus Dexamethasone: Oral netupitant/palonosetron (300 mg/0.50 mg) hard capsule (on Day 1) with oral dexamethasone prior to each scheduled chemotherapy cycle
  Netupitant/Palonosetron
  Dexamethasone
Period: Overall Study
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Started | 203 | 202
Completed | 120 | 117
Not Completed | 83 | 85

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone | Total
Number analyzed (Participants) | 203 | 201 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.7) | 58.9 (10.6) | 59.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 94 | 190
  Male | 107 | 107 | 214
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 201 | 200 | 401
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG performance status [Count of Participants; unit: Participants] — The ECOG Scale is a standard criteria for measuring how the cancer disease impacts a patient's daily living abilities (known to physicians and researchers as a patient's performance status). It describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). There 6 grades, where the performance gets worsening from 0 (patient is fully active, able to carry on all pre-disease performance without restriction) to 5 (patient is dead).
  Participants
    Grade 0 | 81 | 83 | 164
    Grade 1 | 117 | 113 | 230
    Grade 2 | 5 | 5 | 10
Alcohol consumption [Count of Participants; unit: Participants]
  None | 126 | 118 | 244
  Occasional | 76 | 75 | 151
  Regular | 1 | 8 | 9
Tobacco consumption [Count of Participants; unit: Participants]
  Non-smoker | 83 | 77 | 160
  Ex-smoker | 62 | 69 | 131
  Occasional | 0 | 0 | 0
  Regular | 58 | 55 | 113

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Adverse Events
Description: This is a safety study where Adverse Events is the primary outcome (defined by the current ICH Guideline for Good Clinical Practice). Patients are randomized according to a 1:1 ratio (IV NEPA FDC : oral NEPA FDC). No formal comparison is planned, the presence of a control in the same patient population helps interpret any unexpected safety finding in the experimental arm. It is expected that the number of patients randomized to the test group, i.e., 200, will allow approximately 100 patients to be treated with the test drug for 4 cycles. Based on 100 patients treated at Cycle 4 with the IV NEPA FDC , if a given Adverse Event (AE) is not observed, an AE incidence of 3% or greater can be excluded with 95% confidence.
Time Frame: Participants will be followed for the duration of the chemotherapy, an expected average duration of up to 14 weeks assuming a maximum of 4 chemotherapy cycles given every 3 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants
  Any TEAE | 169 | 174
  Severe TEAE | 86 | 90
  Serious TEAE | 41 | 43
  TEAE leading to death | 10 | 14
  TEAE leading to discontinuation from the study | 16 | 20

2. Secondary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication, in the Acute Phase
Time Frame: 0-24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 188 | 182

3. Secondary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication, in the Delayed Phase
Time Frame: >24-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 159 | 176

4. Secondary Outcome: Percentage of Patients With Complete Response (CR) Defined as no Emesis, no Rescue Medication, in the Overall Phase
Time Frame: 0-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 156 | 169

5. Secondary Outcome: Percentage of Patients With no Emetic Episodes in the Acute Phase
Time Frame: 0-24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 164 | 165

6. Secondary Outcome: Percentage of Patients With no Emetic Episodes in the Delayed Phase
Time Frame: >24-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 173 | 184

7. Secondary Outcome: Percentage of Patients With no Emetic Episodes in the Overall Phase
Time Frame: 0-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 171 | 178

8. Secondary Outcome: Percentage of Patients With no Significant Nausea (VAS <25 mm) During the Acute Phase
Time Frame: 0-24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 183 | 187

9. Secondary Outcome: Percentage of Patients With no Significant Nausea (VAS <25 mm) During the Delayed Phase
Time Frame: >24-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 165 | 179

10. Secondary Outcome: Percentage of Patients With no Significant Nausea (VAS <25 mm) During the Overall Phase
Time Frame: 0-120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
Number analyzed (Participants) | 203 | 201
Participants | 161 | 174

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Pro-netupitant/Palonosetron Plus Dexamethasone | Netupitant/Palonosetron Plus Dexamethasone
All-Cause Mortality (participants affected / at risk) | 10/203 | 14/201
Serious Adverse Events (participants affected / at risk) | 41/203 | 43/201
Other Adverse Events (participants affected / at risk) | 169/203 | 174/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pro-netupitant/Palonosetron Plus Dexamethasone (N=203) | Netupitant/Palonosetron Plus Dexamethasone (N=201)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Death (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 1
Sudden death (General disorders) | 1 | 3
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 4
Pyopneumothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 4
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Anuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pro-netupitant/Palonosetron Plus Dexamethasone (N=203) | Netupitant/Palonosetron Plus Dexamethasone (N=201)
Anaemia (Blood and lymphatic system disorders) | 33 | 38
Leukopenia (Blood and lymphatic system disorders) | 21 | 22
Neutropenia (Blood and lymphatic system disorders) | 61 | 58
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 11
Constipation (Gastrointestinal disorders) | 21 | 26
Nausea (Gastrointestinal disorders) | 20 | 14
Asthenia (General disorders) | 13 | 17
Fatigue (General disorders) | 18 | 17
Alanine aminotransferase increased (Investigations) | 15 | 24
Aspartate aminotransferase increased (Investigations) | 12 | 19
Blood creatinine increased (Investigations) | 12 | 6
Decreased appetite (Metabolism and nutrition disorders) | 7 | 11
Headache (Nervous system disorders) | 11 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 32 | 29
Hypertension (Vascular disorders) | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less